CLINICAL TRIAL: NCT07193823
Title: Sexual Dysfunction Prevalence and Its Relationship With Various Factors in Women With Multiple Sclerosis
Brief Title: Sexual Dysfunction in Women With Multiple Sclerosis (MS)
Acronym: MS
Status: Recruiting | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Merve Dokumaci, Resident Doctor, Department of Physical Medicine and Rehabilitation, Ege University
Other Study IDs: 24-5.1T/1
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting; Fatigue in Multiple Sclerosis; Sexual Disfunction; Cognitive Dysfunction; Depression; Anxiety; Overactive Bladder; Fatigue
Keywords: multiple sclerosis; sexual dysfunction; cognitive dysfunction; depression; anxiety; overactive bladder; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Cognitive Dysfunction; Depression; Anxiety Disorders; Urinary Bladder, Overactive; Fatigue; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Sexual dysfunction in women with multiple sclerosis (MS) is an important yet often overlooked problem. The primary objective of this study is to investigate the prevalence of sexual dysfunction in female patients diagnosed with MS. The secondary objective is to evaluate the relationship between sexual dysfunction and fatigue, depression, anxiety, overactive bladder symptoms, and cognitive dysfunction.

For this purpose, the following validated instruments will be used: the Female Sexual Function Index (FSFI) to assess sexual dysfunction, the Brief International Cognitive Assessment for MS (BICAMS) to evaluate cognitive function, the Hospital Anxiety and Depression Scale (HADS) to assess depression and anxiety, the Fatigue Severity Scale (FSS) to measure fatigue, and the Overactive Bladder Questionnaire (OAB-V8) to evaluate overactive bladder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 25-50 years
* Literate and able to comprehend written and spoken instructions
* Diagnosed with relapsing-remitting form of multiple sclerosis
* Having a continuous/regular sexual partner
* Expanded Disability Status Scale (EDSS) score ≤ 5
* At least 3 months since the last relapse
* Sexually active within the past 3 months
* Spasticity level < grade 2 according to the Modified Ashworth Scale

Exclusion Criteria:

* Pregnancy
* Illiteracy or inability to understand spoken or written instructions
* Absence of a continuous/regular sexual partner
* Expanded Disability Status Scale (EDSS) score > 5
* Not sexually active within the past 3 months
* Spasticity level ≥ grade 2 according to the Modified Ashworth Scale

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients with MS under follow-up at the Department of Neurology, Ege University.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sexual dysfunction in female patients with multiple sclerosis | At enrollment (Baseline, cross-sectional assessment)

SECONDARY OUTCOMES:
Association between sexual dysfunction and cognitive dysfunction, fatigue, depression, anxiety, and overactive bladder symptoms | At enrollment (Baseline, cross-sectional assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Akkoc, M.D., Prof, Study Director — Ege University Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Ege University Faculty of Medicine, Department of Neurology, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT07193823/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT07193823/ICF_001.pdf